CLINICAL TRIAL: NCT00969007
Title: Identification of Predictors of Success for Lifestyle Modifications in Overweight Pre-diabetic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marie-France Langlois (Other)
Collaborators: The Lawson Foundation (Other)
Responsible Party: Sponsor-Investigator, Marie-France Langlois, MD, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-083
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Glucose Intolerance; Obesity
MeSH Terms: conditions — Glucose Intolerance; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling (Experimental)
  Interventions: Behavioral: Lifestyle modification counselling

INTERVENTIONS:
Behavioral: Lifestyle modification counselling — Patients meet individually every six weeks, a nurse or kinesiologist, and a dietitian (as well as a psychologist, if needed) and every three months an endocrinologist. A unique patient chart is shared by members of the interdisciplinary team, allowing sharing of the information and avoiding repetitions. Individualized behavioural intervention is proposed and focuses on attainable goals and progressive but sustained small changes in nutrition and physical activity. In addition, the participants have access to 24 weekly group seminars, on different aspects of excess weight and modification of lifestyle, to reinforce behaviour and commitment to lifestyle changes. Our approach meets all criteria suggested for clinical intervention in the 2006 Canadian clinical practice guidelines on the management and prevention of obesity in adults and children.

SUMMARY:
The primary objective of the study is to identify baseline and early predictors of favorable and unfavorable response to lifestyle intervention. As a secondary objective, the investigators would like to validate our questionnaire or other identified predictors as clinical tools to guide us in selection of the most suitable candidates for lifestyle intervention programs. Assuming the same capacity of our questionnaire to predict an absence of weight loss (≥5%) or a loss to follow-up (likelihood ratio for a positive test, LR+ = 9.9), 70 subjects need to be included in this study in order to find a lower limit of the 95% confidence interval above 2.0 for this LR+, which is the limit of an acceptable test. The investigators will enroll participants with pre-diabetes and BMI 27-40 in our program and administer to them at baseline and at 3 months the designed questionnaire, as well as other already well validated questionnaires assessing state of change and readiness to implement diet or exercise modifications.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 27-40 kg/m2
* impaired glucose tolerance, confirmed by an oral glucose tolerance test (OGTT = fasting glucose lower than 7.0 mmol/l and glucose 2 hours post 75g of glucose between 7.8-11.0 mmol/l), or impaired fasting glucose (6.1-6.9 mmol/L)
* 18 years old or more
* Being able to read and give an informed consent

Exclusion Criteria:

* Conditions that affects weight or glucose metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
5% weight loss | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Langlois, Principal Investigator — Université de Sherbrooke; Jean-Patrice Baillargeon, MD, M.Sc., Principal Investigator — Université de Sherbrooke
Locations (1):
- Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada